CLINICAL TRIAL: NCT00674726
Title: Prospective Study on the Difference of Axilar-rectal Temperature in Acute Appendicitis
Brief Title: Study on the Difference of Axilo-rectal Temperature in Appendicitis
Status: Withdrawn | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Principal Investigator, MARCELO A. BELTRAN, M.D., DIGESTIVE SURGEON, Cirujanos la Serena
Other Study IDs: HLS-002-05-08
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Appendicitis; Gastroenteritis
Keywords: appendicitis; gastroenteritis; temperature; fever; acute abdomen; Axilo-rectal temperature in appendicitis; Axilo-rectal temperature in gastroenteritis
MeSH Terms: conditions — Appendicitis; Gastroenteritis; Fever; Abdomen, Acute | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: Patients with acute appendicitis
  Interventions: Other: Observation and measurement of axilo-rectal temperature
- Group II: Patients with acute gastroenteritis
  Interventions: Other: Observation and measurement of axilo-rectal temperature

INTERVENTIONS:
Other: Observation and measurement of axilo-rectal temperature — Measurement of axilo-rectal temperature

SUMMARY:
The investigators are studying prospectively the difference in axilo-rectal temperature in patients with acute appendicitis and using as a control group patients consulting with acute gastroenteritis at our emergency unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute appendicitis
* Patients with acute gastroenteritis
* Patients older than 15 years of age

Exclusion Criteria:

* Other acute abdominal diseases

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting in the emergency unit with acute appendicitis or acute gastroenteritis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The real difference in axilo-rectal temperature in patients with acute appendicitis | 6 hours

SECONDARY OUTCOMES:
The differences in axilo-rectal temperature between patients with acute appendicitis and acute gastroenteritis | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Beltran, M.D., Principal Investigator — Hospital de La Serena
Locations (2):
- Chile (2):
  - Hospital de La Serena - Emergency Unit, La Serena, Coquimbo Region
  - Hospital de La Serena, La Serena, Coquimbo Region